CLINICAL TRIAL: NCT02950662
Title: Effect of Polyether Ether Ketone (PEEK) Housing Verses Metallic Housing of Ball and Socket Attachment on Retention of Mandibular Implant Retained Overdentures: Randomized Clinical Trial
Brief Title: (PEEK) Housing Verses Metallic Housing of Ball and Socket Attachment on Retention of Mandibular Overdenture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Ibrahim Eldesoky Mohamed Elbakry, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: cebd-cu-2016-10-230
Record Dates: First submitted 2016-10-25; First posted 2016-11-01 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Problem With Dentures
MeSH Terms: interventions — Denture, Overlay

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metal housing (Active Comparator): metal housing of ball and socket attachment the intervention will be overdenture
  Interventions: Other: Overdenture
- Peek housing (Active Comparator): Peek housing of ball and socket attachment the intervention will be overdenture
  Interventions: Other: Overdenture

INTERVENTIONS:
Other: Overdenture — Active comparator will be metal housing and peek housing
  Other Names: Implant supported overdenture

SUMMARY:
The aim of this study is to compare the clinical effect of PEEK housing vs. metal housing in terms of retention and patient satisfaction

ELIGIBILITY:
Inclusion Criteria:

1. Patient should be free from any systemic disease that may interfere with dental implants placement and/or osseointegration e.g. uncontrolled diabetes, hypertension, blood diseases, bone diseases, smoking.etc.
2. Patients have completely edentulous upper and lower arches.
3. Patients have healthy mucosa free from any ulceration, inflammation or infections.
4. All patients are free from neuromuscular and temporomandibular joint disorders.
5. Selected patients have normal maxillo-mandibular relationship (Angle class I ridge classification) with adequate inter-arch space and normal tongue size.

Exclusion Criteria:

1. Patients with limited manual dexterity.
2. Patients with Xerostomia, excessive salivation or pathological mucosal changes (e.g. Lichen planus, Leukoplakia…etc.)
3. Pregnant females.
4. Un co-operative patients.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Retention of implant supported overdenture by using digital force meter device | 3 months

IPD SHARING:
Plan to Share IPD: Undecided